CLINICAL TRIAL: NCT03718273
Title: A Phase III Clinical Trial to Compare Ivabradine Versus Digoxin in the Heart Rate Control in Patients With Permanent Atrial Fibrillation Under Treatment With Beta-blockers or Calcium Antagonists.
Brief Title: IvaBRAdine blocK of Funny Current for Heart Rate Control in permanEnt Atrial Fibrillation. (BRAKE-AF Study).
Acronym: BRAKE-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adolfo Fontenla (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Adolfo Fontenla, Adolfo Fontenla, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAKE-AF; 2018-001936-23 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Heart Diseases
Keywords: Ivabradine; Digoxin; Atrial Fibrillation; Heart rate control
MeSH Terms: conditions — Atrial Fibrillation; Heart Diseases | interventions — Ivabradine; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digoxin (Active Comparator): Digoxin 0,25 mg. The initial dose will be based on whether there are factors such as age over 80 years, weight under 60 kg and creatinine clearance <60ml / min,
  Interventions: Drug: Digoxin
- Ivabradine (Experimental): Ivabradine 5 mg, twice a day the first month administered by mouth. If the tolerance is good, the dose will be increased to 7.5 mg on month 2 and will continue until the third month.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg, twice a day the first month administered by mouth. If the tolerance is good, the dose will be increased to 7.5 mg on month 2 and will continue until the third month.
  Patients with 75 or more years of age will receive an initial dose of 2.5 mg / twice a day, which can be increased to 5 mg / twice a day in week 7 and to 7.5 mg in month 1 if the tolerance has been good
  Other Names: Ivabradine 5 mg
  Arms: Ivabradine
Drug: Digoxin — The initial dose will be based on whether there are factors such as age over 80 years, weight less than 60 kg and creatinine clearance <60ml / min, if there is no factor, the oral dose will be 0.25mg / 24h. If there are 2 factors, the dose will be 0.15 mg / 24 h. and if there are 2 or 3 factors, the dose will be 0.10 mg / 24 h.
  Other Names: Digoxin 0,25 mg
  Arms: Digoxin

SUMMARY:
The BRAKE-AF Study is a phase III, randomised, controlled, multicentric, open-label clinical trial to prove the noninferiority of ivabradine versus digoxin in the treatment of permanent atrial fibrillation. The total duration of the study is 3 years, with 24 months of enrolment, treatment and follow-up.

DETAILED DESCRIPTION:
This is a non-commercial, investigator-driven clinical study funded through a public competitive call by Instituto de Salud Carlos III, Spanish Ministry of Economy (PI17/01272).

The study is coordinated by the main investigator from Hospital Universitario 12 de Octubre in Madrid; the sponsorship is performed by Dr. Adolfo Fontenla (Hospital Universitario 12 de Octubre). Several responsibilities are delegated to the Clinical Research Unit (Hospital 12 de Octubre, Madrid, Spain).

The study was planned according to the Good Clinical Practices. BRAKE-AF Study has been approved by the Ethics Committee and Spanish Health Authorities. All participating patients must give written informed consent before any study procedure occur.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Permanent Atrial Fibrillation (AF) at the time of randomization, with no prospect of cardioversion, antiarrhythmic treatment with group I or III drugs, or pulmonary vein ablation.
3. Symptoms attributable to AF associated with the presence of at least one of the following inadequate Heart rate (HR) control criteria:

   1. HR at rest > 110 bpm (on ECG -electrocardiogram- performed in the 14 days prior to inclusion).
   2. HR at rest between 80 and 110 bpm (on ECG performed in the 14 days prior to inclusion) and at least one of the following criteria:

   i. HR in exercise of moderate intensity > 130 bpm (measured in an ergometry or in a Holter-ECG performed in the 60 days prior to inclusion).

   ii. Average daytime HR > 80 bpm (measured on a Holter-ECG performed in the 60 days prior to inclusion).
4. Be receiving treatment with beta-blockers or non-dihydropyridine calcium channel blockers (verapamil or diltiazem) at the maximum dose recommended or tolerated by the patient.
5. Be able to voluntarily give their informed consent.
6. B|ood test carried out in the 6 months prior to inclusion' including: blood count, thyroid hormones and creatinine, in order to rule out secondary causes of poor HR control. The creatinine figure will be used to calculate the creatinine clearance in order to adjust the dose of patients who are randomized to the Digoxin group.
7. Transthoracic echocardiogram to rule out, eg, severe valvular heart disease, hypertrophic cardiomyopathy. The one performed in the year prior to inclusion in the study will be considered acceptable provided that the patient's clinical situation has been stable in that period of time.

Exclusion Criteria:

1. Previous treatment or patients with a known contraindication to Ivabradine or Digoxin or to any excipient of both drugs.
2. Paroxysmal or intermittent complete atrioventricular (AV) block in patients not carrying a pacemaker.
3. Decompensated heart failure requiring inotropic and I or intravenous diuretics in the week prior to randomization or in New York Heart Association (NYHA) functional class IV or on the cardiac transplant waiting list,
4. Acute pericarditis, acute myocarditis or constrictive pericarditis.
5. Obstructive hypertrophic cardiomyopathy.
6. Valvular disease requiring surgical or percutaneous correction.
7. Medical causes that justify poor control of heart rate: fever' anemia, hyperthyroidism, pheochromocytoma' etc.
8. Severe hypotension (blood pressure <90/50 mmHg).
9. Concomitant treatment with potent cytochrome P450 3A4 inhibitors such as azole antifungals (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, oral erythromycin, josamycin, telithromycin) HIV protease inhibitors (nelfinavir, ritonavir) and nefazodone.
10. Severe renal insufficiency (CrCl <30 ml/Kg/min) or in a hemodialysis program.
11. Severe hepatic insufficiency.
12. Major surgery (including cardiac surgery) in the month prior to randomization.
13. Severe concomitant illness that supposes a llfe expectancy of less than one year.
14. Impossibility of carrying out scheduled visits to the protocol.
15. Woman of childbearing age (under 50 years of age, except for those who present a gynecological report that proves the presence of menopause) and women who are breastfeeding.
16. Participation in a clinical trial in the previous 6 months.
17. Patients with acute myocardial infarction or unstable angina.
18. Patient with a recent stroke.
19. Patients with congenital long QT syndrome or treated with drugs that prolong this interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Heart rate reduction. | 3 months
  Reduction of the mean daytime heart rate registered in Holter- electrocardiogram (ECG) after treatment with Ivabradine or Digoxin.
Serious adverse events | 3 months
  Proportion of patients experiencing syncope, severe bradycardia or any serious adverse reaction requiring hospitalization, emergency visit or death of the patient during treatment with Ivabradine or Digoxin.

SECONDARY OUTCOMES:
Reduction in the scale of atrial fibrillation (AF) symptoms according to the European Hearth Rhythm Association (EHRA) Score modified. | Months 1 and 3.
  Percentage of patients who experience a reduction in the scale of atrial fibrillation. symptoms according to the EHRA Score modified.
6 minute walk test (6MWT). | Baseline and after 3 months.
  Increase in meters in the 6MWT.
Quality-of-Life Short Form 36 (SF-36) Health Survey (QoL SF-36) Score. | At baseline and 3 months.
  Increase in the score obtained in global quality of life parameters analyzed by the SF-36 questionnaire.
The Atrial Fibrillation Effect on Quality-of-Life (QoL AFEQT) score. | At baseline and 3 months
  Increase in the score obtained in parameters of quality of life quality of life associated with AF analyzed by the AFEQT questionnaire.
Reduction of the daytime Health rate. | 1 month
  Reduction of the average daytime Heart Rate (HR) recorded in Holter-ECG
Reduction of resting Health Rate. | 1 and 3 months
  Reduction of resting heart rate (HR) recorded on one electrocardiogram (ECG).
Reduction of the maximum heart rate (HR) recorded. | 1 and 3 months
  Reduction of the maximum HR recorded in Holter-ECG
Reduction of the mean HR recorded. | 1 and 3 months
  Reduction of the mean HR in 24 hours recorded in Holter-ECG .
Reduction of the HR delta. | 1 and 3 months
  Reduction of the HR delta (difference between maximum HR and mean HR in 24 hours) recorded in Holter-ECG.
Reduction of HR in moderate exercise. | 3 months
  Reduction of HR in moderate exercise (maximum HR measured by Holter-ECG during the 6-minute walk test.
Percentage of patients with non-severe bradycardia. | 1 and 3 months
  Percentage of patients who experience non-severe bradycardia during the study treatment.
Percentage of patients who experience any adverse reaction. | 1 and 3 months
  Percentage of patients who experience any adverse reaction to the study drugs.
Percentage of patients who voluntarily abandon the study drugs. | 3 months
  Percentage of patients who voluntarily abandon the study drugs.
Proportion of hospitalizations, emergency visits and mortality due to a major cardiovascular event. | 3 months
  Proportion of patients experiencing hospitalizations, emergency visits and mortality due to a major cardiovascular event during treatment with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Fontenla, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre
Locations (10):
- Spain (10):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Virgen de la Salud, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fontenla A, Lopez-Gil M, Tamargo-Menendez J, Matia-Frances R, Salgado-Aranda R, Rey-Blas JR, Miracle-Blanco A, Mejia-Martinez E, Pastor-Fuentes A, Toquero-Ramos J, Arias MA, Montilla I, Gomez de la Camara A, Arribas F; BRAKE-AF investigators. Ivabradine for chronic heart rate control in persistent atrial fibrillation. Design of the BRAKE-AF project. Rev Esp Cardiol (Engl Ed). 2020 May;73(5):368-375. doi: 10.1016/j.rec.2019.09.004. Epub 2019 Oct 17. English, Spanish. PMID 31631048